CLINICAL TRIAL: NCT07091201
Title: The Evaluation of the Validity and Reliability The Foot-taping Test in Children With Cerebral Palsy
Brief Title: Validity and Reliability The Foot-taping Test in Children With Cerebral Palsy
Status: Active, not recruiting | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Erdal Horata, PhD; Assistant Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 2024/02-19
Record Dates: First submitted 2025-07-17; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In spastic cerebral palsy, there are interrelated neuromuscular deficits that can affect ankle joint control, including impaired selective voluntary motor control, muscle weakness, spasticity, and shortened muscle-tendon units. As a result, it is important to assess ankle joint control in children with spastic cerebral palsy. Clinicians need valid, reliable, and practical methods to assess ankle joint control. The aim of this study is to evaluate the validity and reliability of the Foot-taping Test in children with spastic cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy is an umbrella term that refers to a permanent group of movement, posture, and/or motor function disorders caused by a non-progressive lesion or abnormality in the developing immature brain. In spastic cerebral palsy, there are interrelated neuromuscular deficits that can affect ankle joint control, impaired selective voluntary motor control, muscle weakness, spasticity, and shortened muscle-tendon units. As a result, it is important to assess ankle joint control in children with spastic cerebral palsy. Clinicians need valid, reliable, and practical methods to assess ankle joint control. The aim of this study is to evaluate the validity and reliability of the Foot-taping Test in children with spastic cerebral palsy. This study will conduct Department of Orthopedic Prosthesis-Orthosis at Afyonkarahisar Health Sciences University Atatürk Health Services Vocational School. Children aged 6-18 with spastic cerebral palsy (diparetic and hemiparetic) from two different special education institutions in the Aegean Region will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* ≤3 diagnosed with spastic cerebral palsy according to the Gross Motor Function and Classification System
* Be between 6 and 18 years of age
* Be diagnosed with spastic diplegic or spastic hemiplegic cerebral palsy
* Have a GMFCS score ≤3
* Have a Communication Function Classification System (CFCS) score ≤2
* Have a Modified Ashworth Scale (MASH) score ≤3 for lower limb muscles
* Be able to walk 10 metres independently
* Be able to follow verbal commands

Exclusion Criteria:

* The presence of serious hearing, vision or cognitive problems,
* The presence of nerve block injections or orthopaedic surgery within the last 6 months (such as Botox injections or muscle lengthening surgery)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with spastic cerebral palsy from two different Special Education Institutions in the Aegean Region will be included in the study. All participants and their guardians will be informed about the aims of the study and the evaluation procedure. Written informed consent will be obtained from all participants and their guardians before the study. The study will be conducted by the principles of the Helsinki Declaration.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Foot-Taping Test | Two assessors will administer the SAVT to the participants on the first day, two hours apart (first test). The duration of the test is 5 minutes. The retest will be administered 7-10 days after the first test.
  For this test, the participant will be asked to strike the floor as quickly as possible for 10 seconds with each bare foot. The number of times the participant taps their foot on the ground within 10 seconds is recorded. The higher the number of times the participant taps their foot, the better their ankle control.
Active Ankle Range of Motion | Two assessors will administer the SAVT to the participants on the first day, two hours apart (first test). The duration of the test is 10 minutes.
  The participant will be placed supine, and the head of the fibula, lateral malleolus, head of the fifth metatarsal, and base of the fifth metatarsal will be marked. A digital camera will be used to photograph the range of motion of active dorsiflexion and plantar flexion. ImageJ, a software, will be used to measure the ROMs from the images.

CONTACTS AND LOCATIONS:
Overall Officials: ERDAL HORATA, PhD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Department of Orthopedic Prosthesis-Orthosis, Afyonkarahisar Health Sciences University, Atatürk Health Services Vocational School, Afyonkarahisar, Turkey (Türkiye)